CLINICAL TRIAL: NCT00800085
Title: Beta Cell Function in (Pre) Type 1 Diabetes
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: AZ-VUB (Other)
Responsible Party: Principal Investigator, Bart Keymeulen, MD PhD, AZ-VUB
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: KD_BF_01
Record Dates: First submitted 2008-11-28; First posted 2008-12-01 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Type 1 Diabetes
Keywords: first degree relatives of type 1 diabetes patients; hyperglycemic clamp test
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FDR of type 1 diabetes patients receiving glucose 20% (No Intervention): First Degree Relatives of diabetes type 1 patient with a high, intermedian or low risk (accoring to the criteria of the protocol), for developing diabetes type 1.
  Interventions: Drug: glucose 20%

INTERVENTIONS:
Drug: glucose 20% — maintain glycemia at 180 mg/dL till 150 min. after start glucose infusion: with a maintenance dose computed at 5- to 10-minute intervals

SUMMARY:
This study will establish criteria indicating short-term loss of beta cell mass and therefore accelerated progression towards type 1 diabetes.

DETAILED DESCRIPTION:
This study will establish criteria indicating short-term loss of beta cell mass and therefore accelerated progression towards type 1 diabetes. These criteria may help to determine the time point and type of prevention may contribute to the composition of homogeneous groups of study subjects (based on residual beta cell mass, homogeneous risk of beta cell destruction during intervention) and may lead to the identification of functional markers that could be used as surrogate endpoints. This may reduce the number of subjects needed to treat as well as the follow-up time necessary to study significant effects of the test substance.

ELIGIBILITY:
Inclusion Criteria:

* The following groups of first degree relatives of type1 diabetes patients with normal glucose tolerance during OGTT (5-39 years) will be included after informed consent on the basis of their antibody status (n = 40 per group):

  * IA-2A-positives;
  * Ab.-positives (positive for at least 2 different Abs. (IAA, GADA and/or ICA) and/or persistently Ab.-positive for 1 of these Abs;
  * persistently Ab.-negatives.
* 40 type 1 diabetes patients with the following criteria will be studied: 1) aged 12-39 years; 2) < 4 weeks of insulin treatment; 3) auto-Ab.-positive; 4) polyuria since < 6 months; 5) < 10% weight loss over the last 6 months; 6) informed consent.

Exclusion Criteria:

* Pregnancy or lactation in women
* Use of illicit drugs or overconsumption of alcohol (> 3 beers/day) or history of drug or alcohol abuse
* Being legally incapacitated, having significant emotional problems at the time of the study, or having a history of psychiatric disorders
* Having received antidepressant medications during the last 6 months
* Treatment with immune modulating or diabetogenic medication (such as corticosteroids)
* Presently participating in another clinical study
* History of any illness that, in the opinion of the investigator, might confound the results of the study or pose additional risks to the subjects

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-10; Primary Completion 2014-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
The systematic and simultaneous determination of markers of functional beta cell mass and immune status allows stratification according to the stage of the pathogenic process rather than according to a late metabolic consequence of this process | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: katelijn Decochez, MD PhD, Principal Investigator — UZ Brussels
Locations (4):
- Belgium (4):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - UZ Brussels, Brussels
  - UZ Gent, Ghent
  - UZ Leuven, Leuven

REFERENCES:
- [Background] DeFronzo RA, Tobin JD, Andres R. Glucose clamp technique: a method for quantifying insulin secretion and resistance. Am J Physiol. 1979 Sep;237(3):E214-23. doi: 10.1152/ajpendo.1979.237.3.E214. PMID 382871
- [Background] Gorus FK, Goubert P, Semakula C, Vandewalle CL, De Schepper J, Scheen A, Christie MR, Pipeleers DG. IA-2-autoantibodies complement GAD65-autoantibodies in new-onset IDDM patients and help predict impending diabetes in their siblings. The Belgian Diabetes Registry. Diabetologia. 1997 Jan;40(1):95-9. doi: 10.1007/s001250050648. PMID 9028724
- [Background] Decochez K, De Leeuw IH, Keymeulen B, Mathieu C, Rottiers R, Weets I, Vandemeulebroucke E, Truyen I, Kaufman L, Schuit FC, Pipeleers DG, Gorus FK; Belgian Diabetes Registry. IA-2 autoantibodies predict impending type I diabetes in siblings of patients. Diabetologia. 2002 Dec;45(12):1658-66. doi: 10.1007/s00125-002-0949-8. Epub 2002 Nov 12. PMID 12488955
- [Background] Achenbach P, Warncke K, Reiter J, Naserke HE, Williams AJ, Bingley PJ, Bonifacio E, Ziegler AG. Stratification of type 1 diabetes risk on the basis of islet autoantibody characteristics. Diabetes. 2004 Feb;53(2):384-92. doi: 10.2337/diabetes.53.2.384. PMID 14747289
- [Background] Bingley PJ, Gale EA; European Nicotinamide Diabetes Intervention Trial (ENDIT) Group. Progression to type 1 diabetes in islet cell antibody-positive relatives in the European Nicotinamide Diabetes Intervention Trial: the role of additional immune, genetic and metabolic markers of risk. Diabetologia. 2006 May;49(5):881-90. doi: 10.1007/s00125-006-0160-4. Epub 2006 Mar 3. PMID 16514546
- [Background] Maclaren N, Lan M, Coutant R, Schatz D, Silverstein J, Muir A, Clare-Salzer M, She JX, Malone J, Crockett S, Schwartz S, Quattrin T, DeSilva M, Vander Vegt P, Notkins A, Krischer J. Only multiple autoantibodies to islet cells (ICA), insulin, GAD65, IA-2 and IA-2beta predict immune-mediated (Type 1) diabetes in relatives. J Autoimmun. 1999 Jun;12(4):279-87. doi: 10.1006/jaut.1999.0281. PMID 10330299